CLINICAL TRIAL: NCT07328776
Title: A Multi-stage Evaluation Foundation Model for Anti-VEGF Therapy Decision: A Randomized Control Trial
Brief Title: An Assistant Model for Anti-VEGF Therapy Decision
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaodong Sun, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SXD20251227
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Exudative Age-Related Macular Degeneration; DME; Retinal Vein Occlusion (RVO)
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FM-VEGF-CDSS assisted arm (Experimental)
  Interventions: Other: FM-VEGF-CDSS assisted
- without FM-VEGF-CDSS assisted arm (Active Comparator)
  Interventions: Other: without FM-VEGF-CDSS

INTERVENTIONS:
Other: FM-VEGF-CDSS assisted — A Comprehensive Deep Learning Model for Assisting the decision of anti-VEGF therapy: FM-VEGF-CDSS system
  Arms: FM-VEGF-CDSS assisted arm
Other: without FM-VEGF-CDSS — without FM-VEGF-CDSS
  Arms: without FM-VEGF-CDSS assisted arm

SUMMARY:
We present FM-VEGF-CDSS system, the first foundation model-based AI system specifically designed for the decision of anti-VEGF therapy by emulating clinician decision-making reasoning process for those with exudative retinal diseases. FM-VEGF-CDSS is capable of processing multimodal input including optical coherence tomography (OCT) and descriptive medical metadata. Trained and validated on cases from centers across China, the system performed well in both internal and external validation dataset, and could generate the convenient report to enhance decision-making interpretability. To validate its clinical practice, we conducted a prospective multicenter RCT, rigorously assessing FM-VEGF-CDSS system's prediction accuracy and real-world utility. This will improve the standardized decision for anti-VEGF therapy, promoting health equity.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with clinical features suggestive of exudative retinal diseases based on the initial assessment by the physician

Exclusion Criteria:

* Refusal to undergo OCT testing; Refusal to complete the 6-month follow-up period; Screening for a history of intraocular surgery in both eyes within the past 6 months; Subjects with severe systemic diseases, intellectual developmental disorders, psychiatric illnesses, etc.

Patient data that the investigator deems necessary to exclude.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The prediction accuracy of anti-VEGF therapy interval | From enrollment to the end of follow-up at 6 months or to the next anti-VEGF therapy

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Sun, PhD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Shanghai general hospital, Shanghai Jiao Tong University, Shanghai, 200080, Shanghai
  - Shanghai general hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided